CLINICAL TRIAL: NCT02733952
Title: Intravenous Tranexamic Acid Versus Pericervical Tourniquet To Decrease Blood Loss In Trans-Abdominal Myomectomy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Mohamed Bahaa Eldin Ahmed, Clinical professor, Ain Shams Maternity Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ASUObGyn
Record Dates: First submitted 2016-03-27; First posted 2016-04-12 (Estimated); Last update posted 2016-04-12 (Estimated); Status verified 2016-04

CONDITIONS: Post Operative Hemorrhage
MeSH Terms: conditions — Postoperative Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- tranexamic acid (Active Comparator): bolus intravenous injection of tranexamic acid 10mg/kg (maximum1g) 15 min before incision followed by continuous infusion of 1mg/kg/h dissolved in 1L of saline for 10 h (maximum
  1 g/10 h)
  Interventions: Drug: Tranexamic Acid
- Pericervical Tourniquet (Active Comparator): The tourniquet method will be used where the urinary bladder will be dissected downwards from the lower uterine segment, and then a perforation will be made in the posterior leaflet of the broad ligament bilaterally at the level of uterine isthmus. A tourniquet (using 16- inch Foley catheter) will be passed through the perforation encircling the uterine arteries bilaterally. The Fallopian tubes and the ovaries will be carefully excluded from the line of the tourniquet to avoid direct compression and necrosis. The tourniquet will be released intermittently (at about 30 minutes interval) during the surgery and ﬁnally removed after the repair of the uterus
  Interventions: Procedure: Pericervical Tourniquet

INTERVENTIONS:
Drug: Tranexamic Acid
  Other Names: Kapron
  Arms: tranexamic acid
Procedure: Pericervical Tourniquet
  Arms: Pericervical Tourniquet

SUMMARY:
Intravenous Tranexamic Acid Versus Pericervical Tourniquet To Decrease Blood Loss In Trans-Abdominal Myomectomy

DETAILED DESCRIPTION:
this study aims at comparing between different methods to decrease blood loss in trans-abdominal myomectomy. this study compares between medical (intravenous tranexamic acid administration) and non medical (pericervical tourniquet) methods in decreasing blood loss intra operative

ELIGIBILITY:
Inclusion Criteria:

* • Women in the reproductive age (20 - 40 years) diagnosed as having uterine fibroids who are consenting to have trans-abdominal myomectomy in the postmenstrual period diagnosed by:

Clinical symptoms and signs:

* Abnormal uterine bleeding (menorrhagia or (and) metrorrhagia).
* Pain (dull aching lower abdominal pain or dysmenorrhea).
* Pressure symptoms (dyspareunia, dysuria, dyschezia or (and) backache).
* Progressive abdominal enlargement (abdominal swelling).

All women with clinical presentation suggestive of uterine fibroid will undergo abdominal and trans-vaginal ultrasound to confirm the clinical diagnosis and to exclude patients with:

* Submucous uterine myomas.
* Cervical or supracervical myomas.
* Broad ligamentary and pedunculated myomas.
* Associated pelvic pathology.

Ultrasound criteria of uterine fibroids of included patients:

* Maximum diameter of the largest fibroid is greater than 4cm.
* Maximum number of uterine myomas is not to be more than 5 myomas.
* Uterine fibroid may be subserous or intramural.

Exclusion Criteria:

* Obesity (body mass index >30 kg/m2).
* Cardiac, endocrine, pulmonary or hematological disease (including anemia; hemoglobin level below 10gm/dl).
* Patients known to be allergic to tranexamic acid.
* Patients who received pre-operative hormonal therapy (such as a GnRH analogue).
* Patients presented by or with suspected malignant gynecological disease.
* Patients diagnosed as having submucous uterine fibroids, cervical or supracervical fibroids, broad ligamentary fibroids and pedunculated fibroids.
* Patients with contraindication to general anaesthesia.
* Patients with positive pregnancy test.
* Virgin patients.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2015-08; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Estimated intra-operative blood loss measured in milliliters | first 24 hours postoperative

SECONDARY OUTCOMES:
The need for intra-operative blood transfusion | 1 hour
  It is indicated when intra-operative blood loss exceeds 15% of the patient's estimated blood volume, which is equal to the patient's weight in kilograms multiplied by 10
The need for conversion from myomectomy to hysterectomy | 1 hour
  It is indicated when there is uncontrolled intra-operative hemorrhage affecting the patient's vital signs and not responsive to conservative measures or when it is impossible to reconstruct the uterus because of the many defects left by the removal of multiple fibroids
Operative time in minutes | 1 hour
Intra-operative or post-operative complications | 24 hours
Difference between Pre and post-operative hemoglobin and hematocrit levels | 24 hours
  Postoperative hemoglobin and hematocrit levels are to be measured 24 hours after the operation via a venous blood sample).
Duration of hospital stay in days | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Ahmad M BahaaEldin, MD, Principal Investigator — Ain Shams university maternity hospital
Locations (1):
- Ain shams university maternity hospital, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No